CLINICAL TRIAL: NCT06248710
Title: Effects of Intranasal Oxytocin on Trust Towards Therapists and Dogs: A Randomized Controlled Trial in Healthy Adults
Brief Title: Dog Presence and Oxytocin on Trust Towards Therapists
Acronym: DOT
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Dr. Karin Hediger (Other)
Responsible Party: Sponsor-Investigator, Dr. Karin Hediger, Prof. Dr. Karin Hediger, University of Basel
Organization: University of Basel (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2023-00523
Record Dates: First submitted 2024-01-22; First posted 2024-02-08 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Depressive Symptoms; Human-Animal Interaction
Keywords: Depressive Symptoms; Human-Animal Interaction; Animal-Assisted Interventions; Trust
MeSH Terms: conditions — Depression; Human-Animal Interaction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Condition 1: Oxytocin + dog present (Experimental)
  Interventions: Drug: Oxytocin nasal spray; Other: Animal-Assisted Intervention
- Condition 2: Oxytocin + no dog present (Experimental)
  Interventions: Drug: Oxytocin nasal spray
- Condition 3: Placebo + dog present (Experimental)
  Interventions: Other: Animal-Assisted Intervention; Drug: Placebo
- Condition 4: Placebo + no dog present (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin nasal spray — Syntocinon nose spray is usually applied in the context of labour and breast feeding. In this study, however, it will be used to induce an oxytocin (OT) release. Participants will apply three sprays in each nostril which will result in a dose of 24 I.U of oxytocin per participant
  Arms: Condition 1: Oxytocin + dog present; Condition 2: Oxytocin + no dog present
Other: Animal-Assisted Intervention — The dogs involved in the study are trained and used to work with different people in animal-assisted interventions. The dog will be familiarized with the room and the material as well as the staff of the study. The dog will be specifically trained for this study. The dog will be involved for a maximum of 3 sessions per day (approx. 20 minutes in total) and 2 days per week.
  Arms: Condition 1: Oxytocin + dog present; Condition 3: Placebo + dog present
Drug: Placebo — The placebo nose spray contains a saltwater solution and will be applied like the Syntocinon nose spray containing oxytocin.
  Arms: Condition 3: Placebo + dog present; Condition 4: Placebo + no dog present

SUMMARY:
Oxytocin has been proposed as a neuroendocrine mechanism that may mediate the relationship between dog ownership and positive health outcomes and be linked to human-dog interactions and is thought to be a mechanism of interspecies bonding. While the role of oxytocin in human bonding behaviours and social behaviour, in general, is becoming well-established the role of oxytocin in human-animal interaction and Animal-Assisted Interventions (AAI) remains unclear. This research gap calls for more high-quality research investigating this possible neuroendocrine underlying mechanism to advance knowledge about AAI. If oxytocin indeed might be involved in interspecies bonding, intranasally administered oxytocin should not only enhance trust toward a human but also towards a dog.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Signed informed consent

Exclusion Criteria:

* Pregnancy
* Being scared of dogs or dog hair allergy by self-report
* Any acute or chronic disease (e.g., chronic pain, hypertension, heart disease, renal disease, liver disease, diabetes, respiratory disease, skin pathologies etc.)
* Current medications (psychoactive medication, narcotics, intake of analgesics) or being currently in psychological or psychiatric treatment
* Drug consumption (THC, cocaine, heroin, etc.) within the past 24h before study appointment
* Ongoing psychotherapy treatment
* Sexual Intercourse within the past 24h before study appointment
* Current disease involving respiratory system (e.g., influence, asthma etc.)
* Insufficient German language skills to understand the instructions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2024-01-29 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Trust in the therapist | immediately after the intervention
  The main outcome is trust in the therapist, measured by the Trust and Respect Scale.
  The current questionnaire contains 8 items, four for trust and four for respect. Each item is measured on a 7-point Likert scale (1 = "strongly disagree" to 7 = "strongly agree"), of which 4 are formulated negatively. High values indicate high trust toward the therapist for the positively framed items, and for the negatively framed items low values mean high trust toward the therapist.

SECONDARY OUTCOMES:
Trust in the dog | immediately after the intervention
  The secondary outcome "trust in the dog" will be measured with a Visual Analog Scale (VAS).
  The following extremes will be used: no trust to complete trust. High values indicate high trust in the dog.
perceived emotional closeness to the dog | immediately after the intervention
  The Coleman Dog Attitude Scale (C-DAS) is a reliable and validated measure designed to assess attitudes towards dogs.
  The C-DAS is a 24-item self-report measure with an alpha ranging from 0.98 to 0.99.
perceived stress | pre-intervention
  The secondary outcome "perceived stress" will be measured with a Visual Analog Scale (VAS).
  The following extremes will be used: no stress to extreme stress. High values indicate that participants perceive a lot of stress.
perceived stress | immediately after the intervention
  The secondary outcome "perceived stress" will be measured with a Visual Analog Scale (VAS).
  The following extremes will be used: no stress to extreme stress. High values indicate that participants perceive a lot of stress.
level of difficulty | immediately after the intervention
  The secondary outcome "level of difficulty" in talking about a selected stressful event will be measured with a Visual Analog Scale (VAS).
  The following extremes will be used: no difficulty to extreme difficulty. High values indicate that participants find it extremely difficult to talk about a selected stressful event.
therapeutic alliance | immediately after the intervention
  The Therapy Session Questionnaire (in German "Therapiesitzungsbogen für Patienten und Therapeuten") will be used to assess the secondary outcome of "therapeutic alliance".
  The current questionnaire contains 20 items. Each item is measured on a 7-point Likert scale (-3 = "not at all" to +3 = "yes, exactly"). High values indicate high therapeutic alliance.
therapeutic climate | immediately after the intervention
  Therapy Session Questionnaire (in German "Therapiesitzungsbogen für Patienten und Therapeuten") will be used to assess the secondary outcome of "therapeutic climate".
  The current questionnaire contains 20 items. Each item is measured on a 7-point Likert scale (-3 = "not at all" to +3 = "yes, exactly"). High values indicate a good therapeutic climate.
psychological flexibility | pre-intervention
  The secondary outcome "psychological flexibility" will be measured with the psychological flexibility questionnaire (Psy-Flex).
  The Psy-Flex questionnaire consists of six items, which are representative for the six skills. Items are rated on a Likert scale (5 = "very often" to 1 = "very rarely") and are then summed up. Higher scores represent higher psychological flexibility.
psychological flexibility | immediately after the intervention
  The secondary outcome "psychological flexibility" will be measured with the psychological flexibility questionnaire (Psy-Flex).
  The Psy-Flex questionnaire consists of six items, which are representative for the six skills. Items are rated on a Likert scale (5 = "very often" to 1 = "very rarely") and are then summed up. Higher scores represent higher psychological flexibility.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Basel, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
We are planning on sharing the anonymized data on a openly assess platform.

REFERENCES:
- [Background] Algoe SB, Kurtz LE, Grewen K. Oxytocin and Social Bonds: The Role of Oxytocin in Perceptions of Romantic Partners' Bonding Behavior. Psychol Sci. 2017 Dec;28(12):1763-1772. doi: 10.1177/0956797617716922. Epub 2017 Oct 2. PMID 28968183
- [Background] Bakermans-Kranenburg MJ, van I Jzendoorn MH. Sniffing around oxytocin: review and meta-analyses of trials in healthy and clinical groups with implications for pharmacotherapy. Transl Psychiatry. 2013 May 21;3(5):e258. doi: 10.1038/tp.2013.34. PMID 23695233
- [Background] Feldman R, Weller A, Zagoory-Sharon O, Levine A. Evidence for a neuroendocrinological foundation of human affiliation: plasma oxytocin levels across pregnancy and the postpartum period predict mother-infant bonding. Psychol Sci. 2007 Nov;18(11):965-70. doi: 10.1111/j.1467-9280.2007.02010.x. PMID 17958710
- [Background] Kosfeld M, Heinrichs M, Zak PJ, Fischbacher U, Fehr E. Oxytocin increases trust in humans. Nature. 2005 Jun 2;435(7042):673-6. doi: 10.1038/nature03701. PMID 15931222
- [Background] Nagasawa M, Mitsui S, En S, Ohtani N, Ohta M, Sakuma Y, Onaka T, Mogi K, Kikusui T. Social evolution. Oxytocin-gaze positive loop and the coevolution of human-dog bonds. Science. 2015 Apr 17;348(6232):333-6. doi: 10.1126/science.1261022. Epub 2015 Apr 16. PMID 25883356
- [Background] Powell, L., Guastella, A. J., McGreevy, P. D., Bauman, A., Edwards, K. M., & Stamatakis, E. (2018). The physiological function of oxytocin in humans and its acute response to human-dog interactions: A review of the literature. Journal of Veterinary Behavior, 30, 25-32. https://doi.org/10.1016/j.jveb.2018.10.008
- [Background] Crits-Christoph P, Rieger A, Gaines A, Gibbons MBC. Trust and respect in the patient-clinician relationship: preliminary development of a new scale. BMC Psychol. 2019 Dec 30;7(1):91. doi: 10.1186/s40359-019-0347-3. PMID 31888759
- [Background] Coleman, J. A., Green, B., Garthe, R. C., Worthington Jr, E. L., Barker, S. B., & Ingram, K. M. (2016). The Coleman Dog Attitude Scale (C-DAS): development, refinement, validation, and reliability. Applied Animal Behaviour Science, 176, 77-86.
- [Background] Gloster, A. T., Block, V. J., Klotsche, J., Villanueva, J. E., Rinner, M. T. B., Benoy, C., Walter, M., Karekla, M., & Bader, K. (2021). Psy-Flex: A contextually sensitive measure of psychological flexibility. Journal of Contextual Behavioral Science, 22, 13-23. https://doi.org/10.1016/j.jcbs.2021.09.001